CLINICAL TRIAL: NCT00083161
Title: Pilot Study of a Combination of Standard Etoposide/Cisplatin and Metronomic Cyclophosphamide in Patients With Newly Diagnosed Extensive Stage Small Cell Lung Cancer
Brief Title: Cisplatin, Etoposide, and Cyclophosphamide in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gundersen Lutheran Health System (Other)
Responsible Party: Principal Investigator, Ronald Go, Hematologist, Gundersen Lutheran Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000363799; GLO-03-06-06
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Cisplatin; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral cyclophosphamide plus standard cisplatin with etoposide (Experimental): 1. Etoposide 120 mg/m2 IV Days 1-3 or Etoposide 120 mg/ m2 IV Day1 followed by Etoposide 120 mg/ m2 PO BID Days 2-3
  2. Cisplatin 60 mg/m2 IV Day 1 Every 21 days x 4 cycles
  3. Cyclophosphamide 25 mg PO BID Days 8-19 of each cycle
  Interventions: Drug: cisplatin; Drug: cyclophosphamide; Drug: etoposide

INTERVENTIONS:
Drug: cisplatin — 60 mg/m2 IV day 1, every 21 days for 4 cycles.
Drug: cyclophosphamide — 25 mg by mouth BID days 8-19 or each cycle x 4 cycles. After restaging (if no progression) maintenance cyclophosphamide alone 25 mg by mouth BID daily until disease progression
  Other Names: Cytoxan
Drug: etoposide — 120 mg/m2 IV days 1-3 OR 120 mg/m2 IV day 1 and 120 mg/m2 by mouth BID days 2-3
  Other Names: VP-16

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, etoposide, and cyclophosphamide, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cisplatin, etoposide, and cyclophosphamide together works in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of cisplatin, etoposide, and cyclophosphamide in patients with extensive stage small cell lung cancer.
* Determine the effect of this regimen on circulating endothelial cells in the peripheral blood of these patients.

Secondary

* Determine progression-free survival, tumor response rate, and overall survival in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive cisplatin IV over 30 minutes-2 hours on day 1, etoposide IV over 1-2 hours on days 1-3 OR etoposide IV on day 1 and orally twice daily on days 2-3, and oral cyclophosphamide twice daily on days 8-19. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Maintenance therapy: Patients receive oral cyclophosphamide twice daily in the absence of disease progression.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer

  * Extensive stage disease (i.e., disease beyond the hemithorax and cannot be encompassed safely by a tolerable radiation field)
* Measurable disease
* Concurrent CNS metastases allowed provided patient remains asymptomatic

  * Radiotherapy or surgery for uncontrolled symptoms allowed before study entry

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8 g/dL (transfusion allowed)

Hepatic

* ALT ≤ 2 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times ULN

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance ≥ 60 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past year except adequately treated basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Concurrent corticosteroids for brain metastases allowed

Radiotherapy

* See Disease Characteristics
* Prior radiotherapy to any symptomatic site allowed provided the target site(s) was not previously irradiated
* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety | From time of registration to 30 days post treatment of last cycle.
Effect of metronomic chemotherapy on circulating endothelial cells | Baseline to progression
  Collected cycle 1/day 1 of chemotherapy, Cycle 1/day 8, cycle 1/day 22, and then day 85 and 141, and at disease progression.

SECONDARY OUTCOMES:
Progression-free survival | Registration to time of progression
Response rate | From Registration to time of disease progression
Overall survival | From registration to time patient expires

CONTACTS AND LOCATIONS:
Overall Officials: Ronald S. Go, MD, Study Chair — Gundersen Lutheran Center for Cancer and Blood
Locations (1):
- Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin, United States